CLINICAL TRIAL: NCT03407040
Title: Generation of Cancer Antigen-Specific T-cells From Human Induced Pluripotent Stem Cells (iPSC) for Research and Potential Future Therapy
Brief Title: Generation of Cancer Antigen-Specific T-cells From Human Induced Pluripotent Stem Cells (iPSC) for Research and Potential FutureTherapy
Status: Terminated | Type: Observational
Why Stopped: Investigator left NIH
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 180043; 18-C-0043
Record Dates: First submitted 2018-01-20; First posted 2018-01-23 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Gastrointestinal Cancers; Breast Cancer; Pancreatic Cancer; Melanoma; Lung Cancer
Keywords: Blood; Tissue; Immunotherapy; Tumor; Somatic
MeSH Terms: conditions — Gastrointestinal Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Melanoma; Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood lymphocytes, tumor-infiltrating lymphocytes, tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Cancer Patients: Patients with a cancer diagnosis enrolled on protocol 03-C-0277

SUMMARY:
Background:

Researchers want to test if certain cells can be re-programmed into stem cells. Stem cells can keep reproducing for a long time. Cells made by stem cells can be turned into different types of cells. These include cancer-fighting cells, skin cells, etc. The stem cells generated in this study will be used to make specific tumor-fighting cells that can recognize different types of mutations in cancer cells. They may also help identify new tumor mutations that may not have been identified yet.

Objectives:

To test if a certain type of tumor-fighting cells can be re-programmed into stem cells.

Eligibility:

Participants in another Surgery Branch protocol who are at least 16 years old

Design:

Participants already gave samples of blood and/or tumor tissue in the other protocol. They do not need to come back to the clinic or give any other samples.

Participants will give consent for their samples to be used in this study.

Researchers will obtain cells from the samples. They will grow those cells in the lab. They will create stem cells from them.

Researchers will do genetic tests on the samples.

Most tests will not show important health results. But if they do, the participant will be invited to talk to a genetic counselor and get more detailed testing to confirm the results.

Some of the samples and results will be stored indefinitely. They may be used in future research. No personal information will be stored with them.

...

DETAILED DESCRIPTION:
Background:

T-cells are potentially curative for patients with metastatic cancer, but many patients with cancer have T-cells that are terminally differentiated , a condition associated with treatment failure. We have observed that less differentiated T-cells have a greater capacity to proliferate, persist, and destroy large cancer deposits. Advances in regenerative medicine might allow the generation of rejuvenated T-cells from induced pluripotent stem cells (iPSC).

Objectives:

To reprogram patient specimens into induced pluripotent stem cells (iPSC) and differentiate them into different types of somatic cells with the goal to produce cancer antigen-specific T-cells.

To make stored specimens and/or data available to approved research laboratories and investigators.

Eligibility:

Patients enrolled on the National Cancer Institute Surgery Branch (NCI-SB) Cell Harvest protocol 03-C-0277 (Cell Harvest and Preparation for Surgery Branch Adoptive Cell Therapy Protocols).

Patients willing to be consented on this protocol.

Design:

Cells and tissue obtained previously under protocol 03-C-2077.

Reprogramming of cells and tissue into iPSC lines.

Derivation of iPSC lines into T-cells and iPSC progeny capable of supporting T-cell differentiation.

Generation of an iPSC-derived thymic organoid.

Screening of tumor antigen specificity for regenerated T-cells.

In vivo analysis of regenerated T-cells.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with a cancer diagnosis enrolled on protocol 03-C-0277.
* Willing and able to provide informed consent
* Patients must be greater than or equal to 15 years of age.

EXCLUSION CRITERIA:

-Healthy donors enrolled on protocol 03-C-0277.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a cancer diagnosis enrolled on protocol 03-C-0277
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Production of cancer antigen-specific T-cells | Approximately 10 years
  Reprogram patient specimens into induced pluripotent stem cells (iPSC) and differentiate them into different types of somatic cells
Availability of stored specimens and/or data | Approximately 10 years
  Availability of stored specimens and/or data to approved research laboratories and investigators

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nishimura T, Kaneko S, Kawana-Tachikawa A, Tajima Y, Goto H, Zhu D, Nakayama-Hosoya K, Iriguchi S, Uemura Y, Shimizu T, Takayama N, Yamada D, Nishimura K, Ohtaka M, Watanabe N, Takahashi S, Iwamoto A, Koseki H, Nakanishi M, Eto K, Nakauchi H. Generation of rejuvenated antigen-specific T cells by reprogramming to pluripotency and redifferentiation. Cell Stem Cell. 2013 Jan 3;12(1):114-26. doi: 10.1016/j.stem.2012.11.002. PMID 23290140
- [Background] Vizcardo R, Masuda K, Yamada D, Ikawa T, Shimizu K, Fujii S, Koseki H, Kawamoto H. Regeneration of human tumor antigen-specific T cells from iPSCs derived from mature CD8(+) T cells. Cell Stem Cell. 2013 Jan 3;12(1):31-6. doi: 10.1016/j.stem.2012.12.006. PMID 23290135
- [Background] Parent AV, Russ HA, Khan IS, LaFlam TN, Metzger TC, Anderson MS, Hebrok M. Generation of functional thymic epithelium from human embryonic stem cells that supports host T cell development. Cell Stem Cell. 2013 Aug 1;13(2):219-29. doi: 10.1016/j.stem.2013.04.004. Epub 2013 May 16. PMID 23684540
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0043.html